CLINICAL TRIAL: NCT01621360
Title: A Randomized Controlled Trial Comparing Arthroscopic Surgery to Conservative Management of Femoroacetabular Impingement
Brief Title: Hip Arthroscopy Versus Conservative Management of Femoroacetabular Impingement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKSMC-2011-01
Record Dates: First submitted 2011-12-19; First posted 2012-06-18 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Femoroacetabular Impingement
Keywords: Randomized controlled trial; Intention to treat
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthroscopic surgery (Active Comparator): Arthroscopic surgery of the hip plus optimized medical management
  Interventions: Procedure: Arthroscopic hip surgery
- Conservative management (Active Comparator): Physical therapy aimed at strengthening and stabilization of the hip and appropriate analgesic and anti-inflammatory medication.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Procedure: Arthroscopic hip surgery — Hip arthroscopy
  Arms: Arthroscopic surgery
Other: Physical therapy — Physical therapy aimed at strengthening and stabilization of the hip and appropriate analgesic and anti-inflammatory medication.
  Arms: Conservative management

SUMMARY:
The objective of this study is to determine if patients with femoroacetabular impingement (FAI) who undergo arthroscopic hip surgery experience similar outcomes at 2 years post-operative with respect to physical function, pain, and health related quality of life, compared to similar patients who receive conservative management, including medication and physiotherapy.

DETAILED DESCRIPTION:
Arthroscopic surgery is now commonly used to treat patients with femoroacetabular impingement (FAI) however there is a lack of scientific evidence to support its efficacy. Two distinct types of FAI have been defined: cam impingement and pincer impingement. Cam impingement is described as an abnormally prominent anterolateral femoral head-neck junction that rubs against the acetabular rim during flexion resulting in impingement of the acetabular labrum. Pincer impingement is described as an anatomical overcoverage of the femoral head by the acetabulum that impinges the labrum leading to proliferation, or an increase in the prominence of the acetabular rim, further exacerbating the impingement. Previous studies investigating the efficacy of arthroscopic surgery of the knee and shoulder have shown no benefit compared to sham surgery and non-surgical management, therefore strong scientific evidence is needed to support its use in the treatment of hip pathology.

ELIGIBILITY:
Inclusion Criteria:

* patients with femoroacetabular impingement of the hip
* 18 years of age or older
* grade 1, 2 or 3 radiographic severity of osteoarthritis as defined by the Tonnis classification scale.

Exclusion Criteria:

* identified isolated labral tear
* inflammatory or post-infectious arthritis
* previous arthroscopic treatment for hip osteoarthritis
* previous major hip trauma
* Tönnis grade 4 osteoarthritis in two compartments in persons over 60 years of age.
* patients with a major neurologic deficit, serious medical illness (life expectancy less than 2 years or high intraoperative risk) or those who are unable to provide informed consent or who are deemed unlikely to comply with follow-up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Hip Outcome Score (HOS) | 24 months
  The HOS is a disease-specific questionnaire with high reliability and internal consistency. The index has 2 subscales: Activities of Daily Living (ADL) and Sports. Items are scored from 0-4, or N/A which removes item from scoring. The highest potential score is the total number of items with a response multiplied by 4. The item score divided by the highest potential score, multiplied by 100, generates a percentage. A higher score represents a higher level of physical function. The minimal clinically important difference is 9 points for the ADL subscale and 6 points for the Sports subscale.

SECONDARY OUTCOMES:
Non-Arthritic Hip Score | 2 weeks, and at months 3, 6, 12, 18, and 24.
  The Non-Arthritic Hip Score (NAHS) is a validated disease-specific questionnaire, consisting of 20 questions, divided into four domains: Pain, Symptoms, Physical Function, and Participation. Items are scored from 0-4, and added together for an overall total score. A higher score represents a higher level of physical function and less pain and symptoms. The NAHS has demonstrated good validity and has high internal consistency.
Modified Harris Hip Score | 2 weeks, and at months 3, 6, 12, 18, and 24.
  The Modified Harris Hip Score is a modification of the Harris Hip Score which was originally developed for use in total hip arthroplasty patients. The modified version includes only the pain and function domains (range of motion and deformity domains from original version are removed) for a total score out of 100 points, with a higher score indicating greater function and less pain.
SF-12 | 2 weeks, and at months 3, 6, 12, 18, and 24.
  The SF-12 is a 12-item generic general health instrument that evaluates eight domains including restrictions or limitations on physical and social activities, normal activities and responsibilities of daily living, pain, mental health and well-being, and perceptions of health. The SF-12 has been extensively used, and has been shown to be valid, reliable, and responsive in a wide variety of populations and contexts including patients with orthopedic conditions. It is generally accepted that the minimally important difference for the SF-12 ranges from 3-5 points.
Range of Motion | 2 weeks, and at months 3, 6, 12, 18, and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Naudie, MD, FRCSC, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Center, University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Moseley JB, O'Malley K, Petersen NJ, Menke TJ, Brody BA, Kuykendall DH, Hollingsworth JC, Ashton CM, Wray NP. A controlled trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2002 Jul 11;347(2):81-8. doi: 10.1056/NEJMoa013259. PMID 12110735
- [Background] Kirkley A, Birmingham TB, Litchfield RB, Giffin JR, Willits KR, Wong CJ, Feagan BG, Donner A, Griffin SH, D'Ascanio LM, Pope JE, Fowler PJ. A randomized trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2008 Sep 11;359(11):1097-107. doi: 10.1056/NEJMoa0708333. PMID 18784099
- [Background] Neer CS 2nd. Anterior acromioplasty for the chronic impingement syndrome in the shoulder: a preliminary report. J Bone Joint Surg Am. 1972 Jan;54(1):41-50. No abstract available. PMID 5054450
- [Background] Liotard JP, Cochard P, Walch G. Critical analysis of the supraspinatus outlet view: rationale for a standard scapular Y-view. J Shoulder Elbow Surg. 1998 Mar-Apr;7(2):134-9. doi: 10.1016/s1058-2746(98)90223-3. PMID 9593091
- [Background] Gerber C, Terrier F, Ganz R. The role of the coracoid process in the chronic impingement syndrome. J Bone Joint Surg Br. 1985 Nov;67(5):703-8. doi: 10.1302/0301-620X.67B5.4055864.
- [Background] Anderson K, Bowen MK. Spur reformation after arthroscopic acromioplasty. Arthroscopy. 1999 Oct;15(7):788-91. doi: 10.1016/s0749-8063(99)70018-6. PMID 10524832
- [Background] Thompson WO, Debski RE, Boardman ND 3rd, Taskiran E, Warner JJ, Fu FH, Woo SL. A biomechanical analysis of rotator cuff deficiency in a cadaveric model. Am J Sports Med. 1996 May-Jun;24(3):286-92. doi: 10.1177/036354659602400307. PMID 8734877
- [Background] Wuelker N, Plitz W, Roetman B, Wirth CJ. Function of the supraspinatus muscle. Abduction of the humerus studied in cadavers. Acta Orthop Scand. 1994 Aug;65(4):442-6. doi: 10.3109/17453679408995490. PMID 7976295
- [Background] Gosvig KK, Jacobsen S, Sonne-Holm S, Gebuhr P. The prevalence of cam-type deformity of the hip joint: a survey of 4151 subjects of the Copenhagen Osteoarthritis Study. Acta Radiol. 2008 May;49(4):436-41. doi: 10.1080/02841850801935567. PMID 18415788
- [Background] Kassarjian A, Yoon LS, Belzile E, Connolly SA, Millis MB, Palmer WE. Triad of MR arthrographic findings in patients with cam-type femoroacetabular impingement. Radiology. 2005 Aug;236(2):588-92. doi: 10.1148/radiol.2362041987. Epub 2005 Jun 21. PMID 15972331
- [Background] Martin RL, Sekiya JK. The interrater reliability of 4 clinical tests used to assess individuals with musculoskeletal hip pain. J Orthop Sports Phys Ther. 2008 Feb;38(2):71-7. doi: 10.2519/jospt.2008.2677. Epub 2007 Sep 21. PMID 18560194
- [Background] Notzli HP, Wyss TF, Stoecklin CH, Schmid MR, Treiber K, Hodler J. The contour of the femoral head-neck junction as a predictor for the risk of anterior impingement. J Bone Joint Surg Br. 2002 May;84(4):556-60. doi: 10.1302/0301-620x.84b4.12014. PMID 12043778
- [Background] Pfirrmann CW, Mengiardi B, Dora C, Kalberer F, Zanetti M, Hodler J. Cam and pincer femoroacetabular impingement: characteristic MR arthrographic findings in 50 patients. Radiology. 2006 Sep;240(3):778-85. doi: 10.1148/radiol.2403050767. Epub 2006 Jul 20. PMID 16857978
- [Background] Peters CL, Erickson JA. Treatment of femoro-acetabular impingement with surgical dislocation and debridement in young adults. J Bone Joint Surg Am. 2006 Aug;88(8):1735-41. doi: 10.2106/JBJS.E.00514. PMID 16882895
- [Background] Reynolds D, Lucas J, Klaue K. Retroversion of the acetabulum. A cause of hip pain. J Bone Joint Surg Br. 1999 Mar;81(2):281-8. doi: 10.1302/0301-620x.81b2.8291. PMID 10204935
- [Background] Kim YJ, Bixby S, Mamisch TC, Clohisy JC, Carlisle JC. Imaging structural abnormalities in the hip joint: instability and impingement as a cause of osteoarthritis. Semin Musculoskelet Radiol. 2008 Dec;12(4):334-45. doi: 10.1055/s-0028-1100640. Epub 2008 Nov 18. PMID 19016396